CLINICAL TRIAL: NCT00002218
Title: A Phase I Maximum Tolerated Dose Study of CI-1012 in Late-Stage HIV+ Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parke-Davis (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 278B
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-07

CONDITIONS: HIV Infections
Keywords: HIV-1; Dose-Response Relationship, Drug; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: CI-1012

SUMMARY:
To determine the maximum tolerated dose of CI-1012 in late-stage HIV-1-infected patients. To determine the antiretroviral activity of CI-1012 when added to combination therapy. To assess the multiple-dose pharmacokinetic characteristics of CT-1012 when added to combination therapy. To assess the effect of CI-1012 on the pharmacokinetics of other antiretroviral agents.

DETAILED DESCRIPTION:
Doses are escalated based on safety assessments: As soon as a dose meets the criteria for "tolerated" or "not tolerated", doses are escalated or terminated, respectively. All patients are treated for 2 weeks, with follow-up visits scheduled 1 week and 1 month post-treatment.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Serological evidence of late-stage HIV-1 infection (ELISA and Western Blot).
* CD4 T cell count less than or equal to 200 mm3.
* HIV-1 RNA greater than or equal to 5,000 copies/mL.

Exclusion Criteria

Prior Medication:

Excluded:

* Anti-HIV treatment within 8 weeks prior to entry.
* Systemic steroids within 4 weeks prior to entry.

Prior Treatment:

Excluded:

Treatment with anticancer agents within 4 weeks prior to study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - ViRx Inc, Palm Springs, California
  - ViRx Inc, San Francisco, California
  - Central Florida Research Initiative, Maitland, Florida
  - Natl Institutes of Health, Bethesda, Maryland
  - Univ of Michigan, Ann Arbor, Michigan
  - Univ of Utah Med School / Clinical Trials Ctr, Salt Lake City, Utah